CLINICAL TRIAL: NCT01283204
Title: Randomized Phase II Trial of 4-regimen (SP, FL/Tax, FL/Doc, FOLFOX) in Patients With Recurrent or Metastatic Gastric Cancer
Brief Title: Trial of 4-regimen (SP, FL/Tax, FL/Doc, FOLFOX) in Patients With Recurrent or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0596
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Recurrent or Metastatic Gastric Cancer
MeSH Terms: conditions — Recurrence; Stomach Neoplasms | interventions — titanium silicide; Cisplatin; Paclitaxel; Leucovorin; Fluorouracil; Docetaxel; Folfox protocol; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SP(S-1 with cisplatin) (Active Comparator): SP <Every 3 weeks>
  1. Day 1~14 : TS-1 80mg/m2/day (PO)
  2. Day 1 : CDDP 60mg/m2/day IVF 2hours
  3. Day 15~21 : Rest
  Interventions: Drug: SP
- FL/Tax(Paclitaxel with Leucovorin with 5-FU) (Active Comparator): FL/Tax <Every q 3 weeks>
  1. Day1 : Paclitaxel 175mg/m2 IVF for 2hours
  2. Day1 : Leucovorin 20mg/m2 IVF for 1hour
  3. Day1~3 : 5-FU 1000mg/m2 IVF for 24hours
  Interventions: Drug: FL/Tax
- FL/Doc(Decetaxel with Leucovorin with 5-FU) (Active Comparator): FL/Doc <Every q 3 weeks>
  1. Day1 : Docetaxel 75mg/m2 IVF for 1hour
  2. Day1 : Leucovorin 20mg/m2 IVF for 1hour
  3. Day1~3 : 5-FU 1000mg/m2 IVF for 24hours
  Interventions: Drug: FL/Doc
- FOLFOX(Oxaliplatin with Leucovorin with 5-FU) (Active Comparator): FOLFOX <Every q 2 weeks> D1 : Oxaliplatin 100mg/m2 IVF for 2hours D1 : Leucovorin 20mg/m2 IVF for 1hour D1 : 5-FU 400mg/m2 IV bolus D1~2 : 5-FU 1200mg/m2 IVF for 24hours
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: SP — <Every 3 weeks>
  1. Day 1~14 : TS-1 80mg/m2/day (PO),
  2. Day 1 : CDDP 60mg/m2/day IVF 2hours,
  3. Day 15~21 : Rest.
  Other Names: TS-1® with Cisplatin
  Arms: SP(S-1 with cisplatin)
Drug: FL/Tax — <Every q 3 weeks>
  1. Day1 : Paclitaxel 175mg/m2 IVF for 2hours
  2. Day1 : Leucovorin 20mg/m2 IVF for 1hour
  3. Day1~3 : 5-FU 1000mg/m2 IVF for 24hours
  Other Names: Paclitaxel with Leucovorin with 5-FU
  Arms: FL/Tax(Paclitaxel with Leucovorin with 5-FU)
Drug: FL/Doc — <Every q 3 weeks>
  1. Day1 : Docetaxel 75mg/m2 IVF for 1hour
  2. Day1 : Leucovorin 20mg/m2 IVF for 1hour
  3. Day1~3 : 5-FU 1000mg/m2 IVF for 24hours
  Other Names: Docetaxel with Leucovorin with 5-FU
  Arms: FL/Doc(Decetaxel with Leucovorin with 5-FU)
Drug: FOLFOX — <Every q 2 weeks> D1 : Oxaliplatin 100mg/m2 IVF for 2hours D1 : Leucovorin 20mg/m2 IVF for 1hour D1 : 5-FU 400mg/m2 IV bolus D1~2 : 5-FU 1200mg/m2 IVF for 24hours
  Other Names: Oxaliplatin with Leucovorin with 5-FU
  Arms: FOLFOX(Oxaliplatin with Leucovorin with 5-FU)

SUMMARY:
This study is to evaluate the antitumor activity (i.e. progression free survival, overall survival, response rate, etc), safety and quality of life in patient with recurrent or metastatic gastric cancer during 4-regimen (i.e. SP, FL/Tax, FL/Doc, FOLFOX) based chemotherapy. In addition, it is to evaluate efficacy and adverse events of anticancer agents according to the results of pharmacogenetic study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach
* Unresectable metastatic disease or recurred AGC
* Age ≥ 20 years old
* Eastern Cooperative Oncology Group performance status 0-2
* Estimated life expectancy > 12weeks
* Patients with pre-treatment(radiotherapy, chemotherapy) is not carried out. (However, adjuvant chemotherapy using one kind of medication is allowed. It must passed more than 6 months since end of the treatment.) Conventional radiation therapy should be performed before more than 2 weeks. And it is not allowed radiation therapy on primary tumor, measurable lesions, and abdominal
* According to RECIST ver.1.1, using imaging techniques (CT or MRI), measurement possible disease or not measurable, but assessable disease
* Screening laboratory values within the following limits : Hemoglobin ≥ 9 g/dL, Absolute neutrophil count ≥ 1.5 x 10³/L, Platelet count ≥ 75 x 10³/L, Serum creatinine ≤ 1.5 x UNL, Creatinine clearance ≥ 50 mL/min, AST/ALT ≤ 5.0 x UNL
* The patient or protector have to sign a consent form. And he should be able to understand the right to withdraw consent without disadvantage.

Exclusion Criteria:

* Prior chemotherapy (however, previous (neo-)adjuvant chemotherapy allowed if finished at least 6month ago except S-1, Paclitaxel, Docetaxel, Oxaliplatin . Allowed 5-FU, Cisplatin if finished 6month ago)
* Patients with oral intake is impossible or with malabsorption syndrome
* Patients with medically uncontrolled severe complications or infection
* Patients who have central nervous system disorders, mental disorders, or evidence of CNS metastases
* Patient with diagnosed active overlapping cancer within the past 5years except adequately treated carcinoma insitu of the cervix, basal or squamous cell carcinoma of skin
* The possibility(will) of pregnancy , or pregnant and lactating women
* Patients with clinically significant heart disease
* Progression of gastric lesions is not possible to evaluate
* During clinical trials, patient receiving of systemic chemotherapy or other clinical trials drugs or radiotherapy (However, it is possible that palliative radiotherapy treatment for pain relief on primary lesion after more than 2 weeks)
* Peripheral neuropathy of Grade 2 or greater.
* Patients who taking drugs to change of pharmacological activity of S-1 medicine(Warfarin, phenytoin, allopurinol etc.). Except regular treatment of corticosteroids(or equivalent drugs). However, it is allowed the purposes for pre-treatment of study drugs and the control of nausea and vomiting. (However, it is allowed the treatment for acute allergic reactions, or the treatment with low doses (methylprednisolone 20mg or less, or the equivalent drug) from about 6 months)
* Other cases

  * Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety.
  * Psychological condition or dementia that would not permit the subject to complete the study or sign informed consent
  * Patients with dropout sure in clinical trials or cannot be regular follow-up following reasons. For example, psychological, social, family, geographic reasons or a difficult condition of compliance with clinical trial and proper follow up.
  * Poorly controlled chronic liver disease or diabetes mellitus
  * Else, in the investigator's opinion, should exclude the patient from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-03-09; Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
progression free survival(PFS) | 6 weeks
  Imaging assessments will be performed every 6 weeks until radiographically documented PD(Progressive Disease).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea